## University of California, San Diego Consent to Act as a Research Subject

## Beyond Benefits of Q10: Mitochondrial Cocktail for Gulf War Illness

Who is conducting the study, why you have been asked to participate, how you were selected, and what is the approximate number of participants in the study?

Beatrice A. Golomb, MD, PhD is conducting a pilot research study to gather information to aid in the development of a full trial of a cocktail of nutritional supplements that might help reduce symptoms of Gulf War illness in Gulf War veterans who participated in the 1990-91 Persian Gulf War Conflict. You have been asked to participate in this study because you are a Gulf War veteran, deployed to the Middle East between August 1, 1990 and July 31, 1991, and meet symptom criteria for Gulf War illness. Up to 50 participants may be enrolled in this study. This research is funded by the Department of Defense.

New UC San Diego policy may require participants for this study to undergo a COVID test 72 hours prior to each of their study visits. The COVID test will be charged to your insurance and as a result, insured participants may encounter a ~\$10 co-pay. If you do not have health insurance, the cost of the COVID test will be covered by the Cares Act. We will be compensating all participants with an additional \$15 in cash to account for any potential fees.

If your COVID test is negative, the study visit will continue as planned. If your COVID test is positive, the study visit will be rescheduled to a further date.

Why is this study being done?

The purpose of this study is to gather information to enable the successful design and conduct of a large clinical trial which will assess if a specialized compound of multiple nutritional supplements is helpful in reducing the symptoms of Gulf War illness. Determining the number to enroll in a larger study requires information on the magnitude of benefit, and how much that magnitude varies among affected veterans.

What will happen to you in this study and which procedures are standard of care and which are experimental?

## If you agree to be in this study, the following will happen to you:

1. <u>Study Visits</u>: You will be asked to participate in a total of **7 study visits** over a **12 month period**. Study visits will take place at the UC San Diego Altman Clinical and Translational Research Institute (CTRI), 9452 Medical Center Drive La Jolla, CA 92093 and/or your local Quest Diagnostics facility. Some study procedures may be completed remotely through an online Zoom Pro televisit. The visits will look something like this:

| Study Visit Timeline | Study Visit Procedures |
|---|---|
| | Blood Draw, Questionnaires, Exercise Task, Computer games |
| 1. Run-In | |
| | Dispense Run-In study drug |
| 2. Baseline | Blood Draw, Questionnaires, Exercise Task, Computer games, |
| (1-2 weeks after | |
| Run-In) | Randomize and dispense study drug (placebo or active treatment) |

| 3. Month 2 | Blood Draw, Questionnaires, Exercise Task, Computer games |
|---|---|
| 4. Month 6a | Blood Draw, Questionnaires, Exercise Task, Computer games |
| 5. Month 6b<br>(1-2 weeks<br>following 6a visit) | Blood Draw, Questionnaires, Exercise Task, Computer games, Open Label Phase Begins (all participants on active treatment) |
| 6. Month 8.5-9 | Blood Draw, Questionnaires, Exercise Task, Computer games |
| 7. Month 12 | Blood Draw, Questionnaires, Exercise Task, Computer games |

- 2. <u>Physical Assessment</u>: You will have a physical assessment including blood pressure, temperature, heart rate, height, waist circumference, and weight measured.
- 3. <u>Blood Draws/Intravenous Catheter (IV)</u>: **There will be a blood draw per study visit** in order to conduct the assessments to properly adjust the treatment, and you will have up to 750cc (5 tablespoons) of blood drawn. You will be asked to arrive fasting (no food or drink, except for water, for a minimum of 8 hours) prior to each study visit.
  - a. <u>Blood Draw #1</u>: Will occur at the <u>beginning of your visit</u>.
- 4. Questionnaires: You will be asked to complete some questionnaires prior to every study visit about your health history, symptoms, environmental exposures and military service. You may choose to complete some of these questionnaires prior to study visits. You will also be asked to fill out some surveys at home. The home-surveys will be required at least five times during your study participation and involve rating your symptoms daily for one week prior to a study visit.
- 5. <u>Exercise Test</u>: You will participate in a light exercise activity which will involve timed chair rises.
- 6. <u>Computer Games</u>: At each study visit, you will participate in 2 computer games that will test your memory.
- 7. Study Drug: The study drug consists of varying amounts of nutritional supplements including coenzyme Q10, vitamin B<sub>5</sub> (pantothenic acid), vitamin C, vitamin E, L-carnitine, nicotinamide, riboflavin, thiamine, and alpha lipoic acid; or these plus cod liver oil. If you are already taking fish oil/Omega-3s, you will automatically be excluded from the cod liver oil portion of the treatment protocol. During the first 6 months of study participation, you will receive either the active study drug (the nutritional supplement compound) or the placebo (inactive treatment). For the first 6 months of the study, you will have a 50% chance of receiving the active treatment and a 50% chance of receiving the placebo. Neither you nor the study staff will know which treatment you are taking. The study pharmacist will, however, know which treatment you are taking. For the second 6 months of the study, all participants will receive the active treatment. You will be asked to take the study drug (active treatment or placebo) 3 times a day with a meal.

How much time will each study procedure take, what is your total time commitment, and how long will the study last?

The blood draws will take about 10 minutes each. The urine collection will take about 5 minutes. Study questionnaires will take approximately 1.5 hours to complete. The exercise test will take about 5 minutes. The computer games will take up to 60 minutes. The visits will last up to 2-2.5 hours.

What risks are associated with this study?

Participation in this study may involve some added risks or discomforts. These include the following:

- 1. The addition of COVID tests as a potential requirement to participation adds a small burden to the study participant which is greatly outweighed by the benefit of knowing their COVID status.
- 2. Possible bruising, pain, infection or dizziness from the blood draw. All blood draws will be performed by highly-trained nurses, nursing assistants, or phlebotomists to minimize any of these risks. If you have a history of feeling dizzy or faint during a blood draw, please alert our staff and we will do everything possible to make the procedure comfortable for you.
- 3. Stomach discomfort from the study drug. Some people may report stomach upset after taking this nutritional supplement compound. To reduce your risk of stomach discomfort; we suggest that you always take the study drug with a meal.
- 4. Possible fatigue and muscle discomfort from completing the chair rises. If you prefer, you can request a break or stop the testing.
- 5. Loss of confidentiality is a possible risk, but all safeguards will be undertaken to prevent this from happening. Please refer to the confidentiality section below.
- 6. Questionnaires can lead to boredom or annoyance. You can take a break from testing if this occurs. (You are not required to answer any question that makes you uncomfortable; however, all answers are important to the study.)
- 7. We do not anticipate an elevated risk of mood disorders as a result of your participation (and some components of the active treatment have been reported to improve mood). However, if at any point during the study, you are worried about your mood or feel like you may want to harm yourself, please let the study staff know (858-558-4950, x201 or 858-224-2506). A copy of the Mental Health Resource List will be provided to you, which you may refer to for more resources that you can contact.

Because this is a research study, there may be some unknown risks that are currently unforeseeable. You will be informed of any significant new findings.

What are the alternatives to participating in this study? The alternative to participation in this study is to not participate in this study.

What benefits can be reasonably expected?

There may or may not be any direct benefit to you from these procedures. The investigator(s), however, may learn more about Gulf War illness. All participants will receive the opportunity to be

placed on the active treatment (during the open label phase of the study) which may help with their Gulf War illness symptoms.

Can you choose to not participate or withdraw from the study without penalty or loss of benefits? Participation in research is entirely voluntary. You may refuse to participate or withdraw at any time without penalty or loss of benefits to which you are entitled. If you decide that you no longer wish to continue in this study, you will be required to let the study investigator know by calling our office at (858) 558-4950, x201.

You will be told if any important new information is found during the course of this study that may affect your wanting to continue.

Can you be withdrawn from the study without your consent?

You may be withdrawn from the study if you are unable to follow the directions from study staff or Dr. Golomb feels it is in your best medical interest to not participate.

Will you be compensated for participating in this study?

In compensation for your time and travel, you will receive up to \$350 (portioned out to \$50 per study visit), in the form of a Visa Vanilla Gift Card for participating in this research. You will receive the gift card after each study visit.

Are there any costs associated with participating in this study?

You will be required to provide your own transportation to the study visit. Parking will be provided free of cost.

If you are insured, you may encounter a ~\$10 fee as co-pay for the COVID test. However, we have added an additional \$15 to the total compensation to account for this fee. If you get charged more than \$15, please do not hesitate to contact us.

If you are uninsured, you will likely not encounter any fee as you should be covered by the Cares Act. If you do still get charged, please do not hesitate to contact us.

What if you are injured as a direct result of being in this study?

If you are injured as a direct result of participation in this research, the University of California will provide any medical care you need to treat those injuries. The University will not provide any other form of compensation to you if you are injured. You may call the Human Research Protections Program Office at (858) 246-4777 for more information about this, to inquire about your rights as a research subject or to report research-related problems.

What about your confidentiality?

Research records will be kept confidential to the extent allowed by law. Research files are kept in a locked cabinet in a locked room when not in use. The database is on a password-protected computer. Research files and the database will only be accessible to Dr. Golomb and her research team, all of whom have completed confidentiality training. All identifying information will be stored indefinitely.

Department of Defense USAMRMC Human Subjects Protection Office (HRPO) along with the Food and Drug Administration, the Office of Human Research Protections (OHRP) and the

| | e University of California San Diego (UCS eir responsibility to protect human subjects | |
|---|---|---|
| Who can you call if you have question. Dr. Golomb's research staff answered your questions. If you have of Dr. Golomb at (858) 558-4950, x201. | has explained this study to<br>other questions or research-related problem | - |
| <u> </u> | otections Program Office at (858) 246-4777 at your rights as a research subject or to repo | |
| of Rights" to keep. | ent document and a copy of the "Experimen | ntal Subject's Bill |
| You agree to participate. | | |
| Subject's Printed Name | Subject's Signature | Date |
| Person Obtaining Consent's Name | Person Obtaining Consent's Signature | Date |